CLINICAL TRIAL: NCT00771134
Title: Randomised, Double-Blind, Parallel-Group, Placebo-Controlled, Quetiapine-Referenced, Fixed-Dose Study of Lu AA39959 in the Treatment of Depression in Patients With Bipolar I or II Disorder
Brief Title: Efficacy and Safety of Lu AA39959 in Patients With Bipolar Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was previously suspended and is now terminated
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12601A
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Bipolar Disorder
Keywords: Depression; Bipolar I Disorder; Bipolar II Disorder; Placebo-controlled; Double-blind; Randomised controlled; Multicenter; Clinical study; Mania
MeSH Terms: conditions — Bipolar Disorder; Depression; Mania | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lu AA39959 (Experimental)
  Interventions: Drug: Lu AA39959
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Quetiapine (Active Comparator)
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Lu AA39959 — 30mg/day; 15mg B.I.D. for 8 weeks
  Arms: Lu AA39959
Drug: Placebo — B.I.D. for 8 weeks
  Arms: Placebo
Drug: Quetiapine — 300mg/day for 8 weeks
  Other Names: Seroquel
  Arms: Quetiapine

SUMMARY:
This study will evaluate the efficacy and safety of Lu AA39959 in the treatment of depression in patients with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar disorder is a common lifelong psychiatric disorder characterized by recurrent mood swings with manic or hypomanic episodes alternated with depressive episodes of longer duration. Patients spend more time in depression than in (hypo)mania over their life time. The main goals for the treatment of bipolar disorder are resolution of symptoms, return to premorbid level of social functioning and prevention of future episodes.

Although there are many treatments for bipolar disorder, few are approved, and they have limitations in their use due to safety and tolerability issues. Recommendations exist to use mood stabilisers, antipsychotics or a combination thereof with or without antidepressants and the polypharmacy employed in many cases is a reason for concern. There is a major medical need for more effective treatments in monotherapy with a reduced potential for adverse effects. This study evaluates the efficacy and safety of the new drug, Lu AA39959, in treatment of depression in patients with bipolar disorder.

ELIGIBILITY:
Patients suffering from a major depressive episode of bipolar II or I disorder, according to DSM-IV TR

Inclusion Criteria:

* Current major depressive episode of bipolar II or I disorder, according to DSM-IV TR
* Moderate to severe depression
* History of at least one documented mania or hypomania episode
* Absence of current mania or hypomania

Exclusion Criteria:

* Any current psychiatric disorder other than bipolar disorder defined in the DSM-IV TR
* Any substance disorder with the previous 6 months
* Use of any psychoactive medication (including mood stabilizers) within 2 weeks before randomisation and during the study
* ECT within 6 months before the study
* Female of childbearing potential and not using adequate contraception
* Other protocol-defined inclusion and exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms as measured by the change from baseline in total MADRS score | 8 weeks

SECONDARY OUTCOMES:
Global impression (Clinical Global Impression; CGI-BP-Severity/Improvement), depression/anxiety symptoms (Hamilton Depression/Anxiety scale; HAM-D/A), mania symptoms (Young Mania Rating Scale; YMRS), adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- US024, Atlanta, Georgia, United States